CLINICAL TRIAL: NCT06365866
Title: A Phase II Clinical Trial Evaluating the Efficacy of Adding Intraluminal Brachytherapy After Concurrent Chemoradiotherapy (CCRT) for Local-regional Thoracic Esophageal Cancer.
Brief Title: Evaluate the Efficacy of Adding Intraluminal Brachytherapy After CCRT for Local-regional Thoracic Esophageal Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pin-I Huang, Attending Physcian, Division of Radiation Oncology, Department of Oncology, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-06-008B
Record Dates: First submitted 2024-02-26; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Digestive System Diseases; Digestive System Neoplasms; Esophageal Diseases; Neoplasms by Site; Gastrointestinal Diseases; Neoplasms
Keywords: Brachytherapy; Esophageal cancer; External beam radiotherapy; Intraluminal brachytherapy; Survival
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Digestive System Diseases; Digestive System Neoplasms; Esophageal Diseases; Neoplasms by Site; Gastrointestinal Diseases; Neoplasms

STUDY DESIGN:
Intervention Model Description: Add-on treatment to standard treatment (fixed doses allowing dose reduction or dose delay according to the tolerability of individual patients); No control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Add-on of intraluminal brachytherapy with "BRAXX" Esophageal Brachytherapy Applicator. (Experimental): Brachytherapy protocol starts 3 weeks after EBRT (This is "week 1"). After transnasal insertion of the applicator into the esophagus, CT simulation scan(s) with a dummy source in place will be done for further planning procedures, including adjustment of the applicator and 3D treatment planning.
  Interventions: Device: "BRAXX" Esophageal Brachytherapy Applicator.; Radiation: Add-on of intraluminal brachytherapy

INTERVENTIONS:
Device: "BRAXX" Esophageal Brachytherapy Applicator. — The device is intended for use with a commercially available after loader during brachytherapy. The purpose of the device is to deliver a radioactive source to the esophagus. This device is sterile, disposable, and single-use.
Radiation: Add-on of intraluminal brachytherapy — Brachytherapy protocol starts within 12 weeks after EBRT. High-dose-rate (HDR) 5-Gy per fraction is delivered to GTV of esophageal tumor(s), second fraction (if applicable) to be done within 2 weeks after the first fraction, for a total of 5-10Gy in 1-2 fractions will be delivered.

SUMMARY:
The purpose of this study is to observe the safety and effectiveness of the add-on of intraluminal brachytherapy with BRAXX esophageal brachytherapy applicator after definitive CCRT in patients with thoracic esophageal cancer.

DETAILED DESCRIPTION:
Add-on of intraluminal brachytherapy with applicator:

Brachytherapy protocol starts within 12 weeks after EBRT (This is "week 1"). High-dose-rate (HDR) 5-Gy per fraction is delivered to GTV of esophageal tumor(s), second fraction (if applicable) to be done within 2 weeks after the first fraction, for a total of 5-10Gy in 1-2 fractions. GTV coverage D90 should equal 100% of prescription. It is NOT allowed to give concurrent chemotherapy on the days of HDR brachytherapy.

* Prior to undergoing any study-specific procedure, patients must read and sign the current Ethics Committee/Institutional Review Board (IRB)-approved informed consent form. All on-study procedures are permitted within the visit window of ± 2 week. CT with contrast (no contrast if contraindicated) will be done at months 6 and 9; CT or PET/CT will be done at week 12 and month 12; and endoscopy with or without biopsy will be done at week 12, month 6, 9 and 12 for evaluation of tumor response; OPD follows up at week12, month 6, 9 and 12. A patient will be withdrawn from this study in the situation of any grade 4 toxicities. As for any adverse effects≧grade3, dose reduction, or dose delay according to the tolerability of individual patients is allowed. Grade 3 toxicity will cause the rest of the treatment (at least 1 week) until recovery to ≤grade 2 toxicity. If any patient can not tolerate a full course of brachytherapy, the total dose (EBRT+brachytherapy) can be reduced to 60Gy without violation of protocol. The management of adverse effects will follow general principles. Because tumor response is usually observed after completion of treatment, patients will not withdraw from the study because of no response. However, patients should be withdrawn from the study of (1) any grade 4 toxicity or (2) any unexpected cause of SAE that needs to discontinue radiation such as stroke, heart attack, accident, infection, bleeding…etc. Any failure observed during the post-treatment period will be documented, and patients should be withdrawn from the study, facilitating other treatment interventions.
* During this 12-month trial, any other cancer treatment (such as target therapy) and any non-cancer treatment that can increase adverse reactions within the treatment field are prohibited, so as not to affect treatment outcome or cause a change in side effects. The general management of symptoms or other non-cancer-related treatment is allowed, as long as physicians confirm that the interpretation of treatment outcome or side effects will not be influenced.
* The Investigator may use the data collected in this study for future research; which shall be consented by the Subject in the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-85 years, with ECOG performance 0-2.
* Thoracic esophageal cancer with clinical stage I-IV and biopsy proof; patient with stage I-IV cervical esophageal cancer could be recruited in this trial according to Investigator's assessment.
* Complete CCRT with total doses of 45-55Gy to GTV via external beam radiotherapy (EBRT).

Exclusion Criteria:

* According to Investigator's assessment, patients with double cancer or recurrence could be recruited in this trial if they continue to receive systemic therapy.
* Patient with double cancer, esophageal cancer or recurrence who is scheduled for surgery treatment.
* Involvement of tracheal mucosa or bronchial mucosa.
* Stenosis of esophageal lumen that cannot be bypassed by the applicator after EBRT.
* The distribution of the lesions of interest exceeds 10cm range.
* The patient is participating in other clinical trials.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the local control rate at primary tumor site. | 12 months after completion of treatment
  Subjects will be followed every 3 months after treatment, EGD-endoscopy (± biopsy) and PET/ CT scans will be arranged in Months 3, 6, 9, and 12 to evaluate the tumor status.

SECONDARY OUTCOMES:
To estimate overall response rate. | 12 months after completion of treatment
  The overall response rate was observed within 1 year.
To estimate distant metastasis rate. | 12 months after completion of treatment
  Subjects' distant metastasis rate was observed within 1 year.
To estimate progression-free survival rate. | 12 months after completion of treatment
  Subjects' progression-free survival rate was observed within 1 year.
To estimate overall survival status. | 12 months after completion of treatment
  Subjects' overall survival status was observed within 1 year.
To estimate toxicity analysis. | 12 months after completion of treatment
  All toxicities related to the treatment in this clinical trial will be recorded using the Common Toxicity Criteria version 5.0 developed by the National Cancer Institute.
To estimate adverse event. | 3 months after completion of treatment
  Adverse events of less severity are reported on case report forms and submitted with routine data submission. A submission of severe adverse effect (SAE) report includes every admission and ER visit of any reason within 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pin-I Huang, Ph.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan